CLINICAL TRIAL: NCT01700998
Title: Randomized Trial of Magnesium Replacement Therapy to Prevent Acute Renal Failure in Hypomagnesemic Critically Ill Patients
Brief Title: Magnesium Replacement Therapy to Prevent Acute Renal Failure in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Responsible Party: Principal Investigator, Felipe Dal Pizzol, MD, PhD, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MgICU
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Hypomagnesemia
MeSH Terms: interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 250 ml saline 0.9% for 24 hours in an infusion rate solution of 10.4 ml / hr for 3 days repeated during ICU stay if hypomagnesemia occurs.
  Interventions: Drug: Placebo
- Magnesium (Experimental): 48 mEq Magnesium diluted in 250 ml saline 0.9% for 24 hours in an infusion rate solution of 10.4 ml / hr. Therapy is continued for 3 days and repeated if hypomagnesemia occurs during ICU stay
  Interventions: Drug: Magnesium

INTERVENTIONS:
Drug: Magnesium
  Arms: Magnesium
Drug: Placebo
  Arms: Placebo

SUMMARY:
Acute renal failure (ARF) is a serious and common complication in hospitalized patients, occurring in more than 25% of intensive care unit (ICU) patients. Hypomagnesemia is a common disorder, occurring in approximately 12% of hospitalized patients, with an incidence of 60% in ICU patients. The majority of those patients have are asymptomatic hypomagnesemia, and patients with mild hypomagnesemia do not need treatment, only the correction of the underlying cause. Hypomagnesemia potentiates postischemic renal failure in rats, and is associated, in humans, with acute renal failure. To date, there is no study that demonstrated a benefit of maintain normal levels of magnesium in the incidence of ARF in critically ill patients. Thus, we suggest that a treatment aimed to maintain normal magnesium levels during ICU stay can decrease the incidence of ARF. We will perform a randomized clinical trial that will include all patients admitted to an ICU that, develop hypomagnesemia. It will be excluded from the study: patients younger than 18 years, participants from other studies, pregnant women, patients with creatinine greater than or equal to 3.5 mg / dl or on dialysis, patients who used intravenous contrast for radiological studies, patients weighing less than 40kg, suffering from advanced malignant disease, with severe hypomagnesemia (serum magnesium less than or equal to 1.1 mg / dl), with a diagnosis of Torsades de Pointes or symptomatic hypomagnesemia prior to randomization. Patients included in the study will be randomized to one of the following groups: placebo (saline solution 0.9%) or 50% Magnesium Sulfate. Patients will receive an administration of 48 mEq Magnesium diluted in 250 ml saline 0.9% for 24 hours in an infusion rate of 10.4 ml / hr. Therapy will be continued for 3 days, and repeated during ICU stay to maintain magnesium levels in the normal range. Placebo group will receive exactly the same infusion only with saline administration. The therapy will be discontinued if the patient has hypermagnesemia or signs of magnesium intoxication. The main outcome measurement will be the occurrence of ARF during ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* All patients, clinical or surgical, who signed (or their relatives) the informed consent form, which presented hypomagnesemia (with serum magnesium between 1.2 and 1.8 mg / dL), with no symptoms of hypomagnesemia.

Exclusion Criteria:

* Patients younger than 18 years, participants from other studies, pregnant women, patients with admission plasma creatinine greater than or equal to 3.5 mg / dl or on dialysis, patients who used intravenous contrast for radiological studies, patients weighing less than 40kg, patients suffering from advanced cancer, patients with severe hypomagnesemia (serum magnesium less than or equal to 1.1 mg / dl), patients with a diagnosis of Torsades de Pointes or patients with symptomatic hypomagnesemia prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of acute renail failure | During ICU stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
Rate of recovery from ARF | During hospital stay, an expected average of 5 weeks
ICU and hospital length of stay | Hospital discharge, an expected average of 5 weeks
ICU and hospital mortality | Hospital discharge, an expected average of 2 (ICU) and 5 (hospital) weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Ritter, MD, PhD, Study Chair — UNESC
Locations (1):
- Hospital Sao Jose, Criciúma, Santa Catarina, Brazil